CLINICAL TRIAL: NCT04177446
Title: A Multicenter Randomized Controlled Clinical Study With WeiYuan Tai (a Nutritional Supplement) on Nutritional Support of Enhanced Protein in Severe Patients(Tai Shan)
Brief Title: A Study About Nutritional Support of Enhanced Protein in Critical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Yabao Pharmaceutical Group (Industry); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Wei Chen, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-2028
Record Dates: First submitted 2019-10-11; First posted 2019-11-26 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Critical Illness
Keywords: national support; protein; critical illness
MeSH Terms: conditions — Critical Illness | interventions — maltodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Patients will be given basic energy intake according to their weight, and will be extra maltodextrin as the placebo
  Interventions: Dietary Supplement: basic energy intake; Dietary Supplement: maltodextrin
- intervention group (Experimental): Patients will be given basic energy intake according to their weight, and will be extra protein intake
  Interventions: Dietary Supplement: a production consist of various oligopeptides and the whey protein; Dietary Supplement: basic energy intake

INTERVENTIONS:
Dietary Supplement: a production consist of various oligopeptides and the whey protein — patients will be given extra protein intake except the basic energy intake
  Arms: intervention group
Dietary Supplement: basic energy intake — supplement as basic energy intake
Dietary Supplement: maltodextrin — used as placebo in the control group
  Arms: control group

SUMMARY:
This is a prospective randomized controlled trial. 180 patients with critical illness will be included and randomly divided into two groups. In the control group, patients will be fed with basic energy; and in the experiment group, the patients will be given extra protein intake except the basic energy intake. The intervention duration will last 6 days. The primary outcomes of this study are urea nitrogen of 24h and prealbumin(PA). And other outcomes include nutritional status, safety indicators and clinical indicators.

DETAILED DESCRIPTION:
Critical illness patients are commonly in the risk of malnutrition, because of various factors. And nutritional supplement, particularly the supplement of protein, can decrease the nitrogen balance, improve the nutritional status, accelerate the speed of healing and decrease the mortality rate. This is a multi center prospective randomized controlled trial. 180 patients with critical illness will be included and randomly divided into two groups. In the control group, patients will be fed with basic energy; and in the experiment group, the patients will be given extra protein intake except the basic energy intake. The intervention duration will last 6 days. The primary outcomes of this study are urea nitrogen of 24h and prealbumin(PA). And other outcomes include nutritional status(total protein, albumin, grip and calf circumference), safety indicators(liver function, kidney function, tolerance, etc.) and clinical indicators(overall complication rate, length of hospital stay and cost).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as critical illness, stayed in ICU;
2. score of M-nutric ≥ 5;
3. score of 3. APACHE Ⅱ >12;
4. anticipation of length of hospital stay > 6 days;
5. 18 ≤ age ≤ 45;
6. pattens volunteer to attend this study and sigh the inform consent form;

Exclusion Criteria:

1. liver function(AST/ALT) of blood test ≥ 2.5 ULN(upper limit of normal); renal function of blood test > 1.6 ULN;
2. the patients are used or are planned to use the Human Albumin solution within 3 days before receiving enteral nutrition;
3. consume any natural food or something made by natural food;
4. patients are used or are planned to use all-in-one solution or amino acid solution within 3 days before receiving enteral nutrition;
5. anticipation of survival time is less than 5 days;
6. have the contraindications of enteral nutrition;
7. patients are allergic to material of the production;
8. patients who are considered not suitable for this study by investigators;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12-25 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
urea nitrogen of 24h | day6
  the total amount of urea nitrogen in 24 hours
prealbumin(PA) | day6
  the level of prealbumin in blood

SECONDARY OUTCOMES:
total protein | day6
  the total protein level in blood
albumin | day6
  the level of albumin in blood
calf circumference | change from baseline calf circumference at 6 days
  the perimeter of calf
grip | change from baseline grip at 6 days
  the strength(force measured kilograms) of the right hand measured by a hand-held dynamometer (if the right hand is not impossible, the left is ok )
overall complication rate | from the day receiving enteral nutrition to day6
  the over complication rate after receiving enteral nutrition
length of hospital stay | from date of admission in the hospital until the date of discharge, up to 1 year
  the overall time stay in hospital
cost in hospital | from date of admission in the hospital until the date of discharge, up to 1 year
  all the money paid in the hospital
liver function | day6
  the level of AST/ALT in blood
renal function | day6
  the level of creatinine in blood

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Yes
The following data will be shared at the end of the study: demographic data, other baseline data of patients and date of outcomes collected at this research
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data is expected to be available after, December, 2020 and can be used forever
Access Criteria: The information should be used for academic research, medical communication, etc., and is prohibited from being used for commercial gain.

REFERENCES:
- [Result] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Result] Arabi YM, Al-Dorzi HM, Mehta S, Tamim HM, Haddad SH, Jones G, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L, Kumar A, Bagshaw SM, Aldawood AS; PermiT Trial Group. Association of protein intake with the outcomes of critically ill patients: a post hoc analysis of the PermiT trial. Am J Clin Nutr. 2018 Nov 1;108(5):988-996. doi: 10.1093/ajcn/nqy189. PMID 30475959